CLINICAL TRIAL: NCT01843491
Title: A Phase I Clinical Trial Immunizing Healthy Adults With the NMRC-M3V-Ad-PfCA Vaccine to Generate Biologic Reagents for Refining Immunologic Assays Supporting the Development of the Protective Malaria Vaccine NMRC-M3V-D/Ad-PfCA (AdBa)
Brief Title: A Phase I Clinical Trial Immunizing Healthy Adults With the NMRC-M3V-Ad-PfCA Vaccine to Generate Biologic Reagents
Acronym: AdBa
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not go forward with study.
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRC.2012.0006
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ad-PfCA (Experimental): Single injection of Ad-PfCA containing 2 x 10^10 pu total dose in 1 ml of Final Formulation Buffer by intramuscular injection
  Interventions: Biological: Ad-PfCA

INTERVENTIONS:
Biological: Ad-PfCA — Vaccine
  Other Names: NMRC-M3V-Ad-PfCA

SUMMARY:
This is an open label Phase 1 study of the Ad-PfCA vaccine designed to 1) provide reagents for the development and refinement of cell-mediated immunoassays for measuring the human immune response to candidate malaria vaccines (especially protective malaria vaccines such as DNA/Ad-PfCA where better assays are needed to identify the correlates of protective immunity) and 2) to provide a repository of antigen-specific PBMCs that can be used as positive and negative controls in cell mediated immunoassays.

DETAILED DESCRIPTION:
This is an open label Phase 1 study of the Ad-PfCA vaccine designed to 1) provide reagents for the development and refinement of cell-mediated immunoassays for measuring the human immune response to candidate malaria vaccines (especially protective malaria vaccines such as DNA/Ad-PfCA where better assays are needed to identify the correlates of protective immunity) and 2) to provide a repository of antigen-specific PBMCs that can be used as positive and negative controls in cell mediated immunoassays. The study group will consist of up to 35 healthy adults aged 18 to 50 years who have been screened to meet inclusion and exclusion criteria.

Subjects will be eligible for participation regardless of baseline adenovirus 5 serostatus. At least 6 subjects will be "malaria naïve", meaning that 1) they have not been the recipient of a malaria vaccine, 2) they have no history of malaria infection or travel to a malaria endemic region within 6 months of first leukapheresis procedure or 60mL blood draw, 3) they have no history of long-term residence (>5 years) in an area known to have significant transmission of P. falciparum, and 4) they have a negative P. falciparum circumsporozoite (PfCSP) ELISpot assay at baseline. (From herein, for simplicity, we refer to PfCSP simply as CSP). The remaining subjects will have no restrictions regarding receipt of malaria vaccines, travel history or baseline CSP ELISpot results. Although it is more difficult to recruit "malaria-naïve" subjects, the inclusion of at least 6 such subjects should provide a more varied array of immune responses; this may be helpful for assay development.

Eligible subjects will receive a single administration of the Ad-PfCA malaria candidate vaccine at a dose of 2 x 1010 pu by intramuscular injection. Approximately 1 month pre-immunization, study subjects will either have a large number of PBMCs collected by means of leukapheresis, or a simple 60 mL blood draw, dependent upon initial pre-screening. Pre-immunization samples designated for the repository do not require large volume sampling of PBMCs. Rather, a 60 mL whole blood draw is sufficient for repository purposes. Thus, subjects will be separated into sub-groups, dependent upon initial pre-screening. Subjects whose samples are designated for the repository will undergo a simple, 60 mL blood draw in lieu of leukapheresis #1 (sub-group A). Samples assigned for assay development will be obtained from sub-group B.

Approximately 1 month post-immunization, study subjects in both sub-groups will have PBMCs collected by means of leukapheresis. Consultation with immunology experts after post-immunization screening will assist to identify those subjects whose samples do not meet assay development or repository needs. In an effort to eliminate unnecessary procedures for subjects, these individuals will not undergo a second leukapheresis, but will return for their safety visit on day 84.

Prior to each leukapheresis/60 mL blood draw, a sample will be tested by CSP-ELISpot and AMA1 ELISpot; the results will be used to categorize samples (see below). Follow up visits will occur 2, 7, 14, 21, and 84 days following immunization. Depending on guidance from the FDA, subjects will then be followed annually by phone, email, or mailings up to five years from the time of immunization per FDA recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant, non-lactating female) 18 - 50 years of age (inclusive)
* Available and willing to participate for duration of study
* Able and willing to provide written informed consent
* Able to complete an Assessment of Understanding with a score of at least 75% correct
* In good general health with no clinically significant health problems as established by medical history, physical exam, and laboratory screening
* Men, and women of childbearing potential must agree to use effective means of birth control from time of enrollment through the duration of the active phase of the study (3 months following immunization)
* Women: Sexually active females, unless surgically sterile or at least one year post-menopausal, must use an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) prior to dosing of study vaccine, and must agree to continue using such precautions for at least 3 months after immunization. Female subjects unable to bear children must have a note from a Primary Care Provider as proof of her documentation (e.g. tubal ligation or hysterectomy) or must be post-menopausal as appropriate by age with at least one year of amenorrhea.
* Men must agree to use of effective means of birth control. If a male subject has had a vasectomy this will be considered an adequate means of birth control.
* Agree to refrain from blood donation for one year after immunization
* Agree not to travel to a malaria endemic region during the active phase of the study
* Good peripheral venous access

Exclusion Criteria:

* Females who are pregnant (positive urine β-HCG) or nursing at screening or plan on becoming pregnant or plan to nurse from time of screening through the duration of the active phase of the study (3 months following immunization)
* Positive HIV, HBsAg or HCV serology
* An abnormal EKG, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* Weight less than 110 pounds
* Use of systemic immunosuppressant pharmacotherapy (inhaled and topical steroids are allowed) within 60 days of scheduled leukapheresis/60 mL blood draw or immunization
* Current significant medical condition (cardiovascular, pulmonary, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination (includes bleeding disorders)
* Plan for surgery between screening visit and second (final) leukapheresis
* Known allergy to any component of the vaccine formulation
* Participation in any study involving another investigational vaccine or drug within 30 days prior to the first scheduled leukapheresis/60 mL blood draw or plan to participate in another investigational vaccine/drug research study during participation in the active phase of this study
* Receipt of immunoglobulin and/or any blood products within 90 days of scheduled leukapheresis/60 mL blood draw or immunization
* Any other significant finding which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the study or compromise the scientific objectives
* Risk factors for HIV exposure: unsafe sex and injectable drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Collection | 26 weeks
  Collection of sufficient PBMCs for the laboratory investigators to determine the accuracy, precision, cell usage, throughput, and cost of each of the developed, expanded, or refined immunological assays
ELISpot assay, flow cytometry assay and HLA typing | 26 weeks
  Collection of sufficient PBMCs to meet the minimum required response for positive controls (250 spot forming cells (sfc)/ million PBMCs), with each positive sample characterized using frozen ELISpot assay, flow cytometry assay and HLA typing
Repository | 26 weeks
  Collection of a sufficient bank of characterized PBMCs that vials can be used as global reference reagents for the standardization of malaria vaccine development-specific cellular immunologic assays worldwide

SECONDARY OUTCOMES:
Safety | 26 weeks
  Occurrence, severity, and duration of any solicited symptoms starting on the day of immunization through Day 7 after immunization
  Occurrence of any unsolicited symptoms, abnormal physical findings, and laboratory values starting from the day of immunization through Day 28 after immunization.
  Occurrence of any serious adverse events, as defined in 21 CFR 312.32, for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Judith Epstein, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Naval Medical Research Center Clinical Trials Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tamminga C, Sedegah M, Regis D, Chuang I, Epstein JE, Spring M, Mendoza-Silveiras J, McGrath S, Maiolatesi S, Reyes S, Steinbeiss V, Fedders C, Smith K, House B, Ganeshan H, Lejano J, Abot E, Banania GJ, Sayo R, Farooq F, Belmonte M, Murphy J, Komisar J, Williams J, Shi M, Brambilla D, Manohar N, Richie NO, Wood C, Limbach K, Patterson NB, Bruder JT, Doolan DL, King CR, Diggs C, Soisson L, Carucci D, Levine G, Dutta S, Hollingdale MR, Ockenhouse CF, Richie TL. Adenovirus-5-vectored P. falciparum vaccine expressing CSP and AMA1. Part B: safety, immunogenicity and protective efficacy of the CSP component. PLoS One. 2011;6(10):e25868. doi: 10.1371/journal.pone.0025868. Epub 2011 Oct 7. PMID 22003411
- [Background] Sedegah M, Tamminga C, McGrath S, House B, Ganeshan H, Lejano J, Abot E, Banania GJ, Sayo R, Farooq F, Belmonte M, Manohar N, Richie NO, Wood C, Long CA, Regis D, Williams FT, Shi M, Chuang I, Spring M, Epstein JE, Mendoza-Silveiras J, Limbach K, Patterson NB, Bruder JT, Doolan DL, King CR, Soisson L, Diggs C, Carucci D, Dutta S, Hollingdale MR, Ockenhouse CF, Richie TL. Adenovirus 5-vectored P. falciparum vaccine expressing CSP and AMA1. Part A: safety and immunogenicity in seronegative adults. PLoS One. 2011;6(10):e24586. doi: 10.1371/journal.pone.0024586. Epub 2011 Oct 7. PMID 22003383